CLINICAL TRIAL: NCT02352454
Title: A Multi-Center, Prospective, Randomized Trial Comparing the Effectiveness of Aurix Therapy to Usual and Customary Care in Venous Leg Ulcers
Brief Title: Effectiveness of Aurix Therapy in Venous Leg Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nuo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM003 Gold
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Venous Leg Ulcers
Keywords: Non Healing Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aurix + UCC (Experimental): Subjects will be treated on average twice a week for the first 2 weeks, and then, once a week thereafter while under active treatment, but actual frequency of treatment will be determined by the treating physician. All subjects will receive Aurix treatment and usual and customary care, which can include advanced therapeutics.
  Interventions: Device: Aurix
- Usual and Customary Care (No Intervention): Subjects will be treated on average twice a week for the first 2 weeks, and then, once a week thereafter while under active treatment, but actual frequency of treatment will be determined by the treating physician. All subjects will receive usual and customary care, which can include advanced therapeutics.

INTERVENTIONS:
Device: Aurix — Aurix is a platelet-rich plasma gel used in the treatment of non-healing wounds. It will be administered twice weekly for 2 weeks then weekly.
  Arms: Aurix + UCC

SUMMARY:
The aim of this trial is to demonstrate the effectiveness of complete wound healing in a prospective, open-label, randomized trial in which venous leg ulcers (VLU)n will be treated using Aurix and compared to patients receiving undefined Usual and Customary Care (UCC)

DETAILED DESCRIPTION:
Recurrence of ulcers in the leg is common; two-thirds of patients are likely to experience recurring ulcers after the first ulcer. While treatment of the underlying venous disease, depending on the mode of treatment, can lower the recurrence rate in many patients, it does not affect recurrence. Aurix is a platelet-rich plasma (PRP) gel used in the treatment of non-healing chronic wounds. The aim of this trial is to demonstrate the effectiveness, measured as complete wound healing, in a prospective, randomized trial in which venous leg ulcers will be treated using Aurix and standard of care and compared 1:1 to patients receiving undefined Usual and Customary Care (UCC).

ELIGIBILITY:
Inclusion Criteria:

1. Medicare eligible
2. ≥18 years of age
3. Proven venous disease
4. The largest non-healing wound, if multiple wounds are present, or the single wound to be treated (Index Ulcer) that is located between and including the knee and the ankle
5. For subjects with potentially multiple eligible VLUs, the largest ulcer will be selected as Index Ulcer for study. There must be at least 4 cm between the Index Ulcer and other ulcers; if all ulcers are closer than 4 cm, the subject should not be enrolled (screen failure)
6. Debrided ulcer size between 2 cm2 and 200 cm2
7. Subject has received UCC care for ≥ 2 weeks at treating wound clinic
8. Demonstrated adequate compression regimen
9. Duration ≥ 1 month at first visit
10. Subject must be willing to comply with the Protocol, which will be assessed by enrolling clinician

Exclusion Criteria:

1. Subjects known to be sensitive to Aurix components (calcium chloride, thrombin, ascorbic acid) and/or materials of bovine origin
2. Presence of another wound that is concurrently treated and might interfere with treatment of index wound by Aurix
3. Ulcer not of VLU pathophysiology (e.g., pure diabetic, vasculitic, radiation, rheumatoid, collagen vascular disease, pressure, or arterial etiology)
4. Patients on chemotherapeutic agents or any malignancy in the wound area
5. Subjects who are cognitively impaired
6. Serum albumin of less than 2.5 g/dL
7. Plasma Platelet count of less than 100 x 109/L
8. Hemoglobin of less than 10.5 g/dL
9. Subject has inadequate venous access for repeated blood draw required for Aurix Administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Time to Heal | 12 weeks
  Aurix plus standard of care versus usual and customary care only. Complete wound closure is defined as skin re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visits 2 weeks apart (FDA Guidance for Industry Chronic Cutaneous Ulcer and Burn Wounds - Developing Products for Treatment, 2006).

SECONDARY OUTCOMES:
Proportion of wounds healed | 12 weeks
  Comparison of proportion of wounds healed over 12 weeks
Change in Quality of Life with Chronic Wounds (W-QOL) Score | 12 weeks
  Change in mean Quality of Life with Chronic Wounds (W-QOL) score between baseline and at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Clausen, PhD, Study Director — Nuo Therapeutics
Locations (23):
- United States (23):
  - Methodist Hospital Wound Care Center, Arcadia, California
  - Beverly Hospital Wound and Hyperbaric Center, Montebello, California
  - Kaweah Delta Rehabiliation Hospital, Visalia, California
  - Bristol Hospital Wound Care Center, Bristol, Connecticut
  - Piedmont, Atlanta, Georgia
  - St. Luke's Wound and Hyperbaric Center, Meridian, Idaho
  - The Center for Wound Healing at FHN, Freeport, Illinois
  - Tufts Medical Center - Center for Wound Healing, Boston, Massachusetts
  - St Joseph Mercy Oakland Hospital Center for Wound Care and Hyperbaric Medicine, Pontiac, Michigan
  - Catskill Regional Medical Center - Wound Healing Center, Harris, New York
  - Orange Regional, Middletown, New York
  - The Wound Center of Niagara, Niagara Falls, New York
  - Onslow Memorial Hospital - Wound Care and Hyperbaric Center, Jacksonville, North Carolina
  - Onslow Memorial Hospital Wound Care and Hyperbaric Center, Jacksonville, North Carolina
  - Berger Wound Healing Center, Circleville, Ohio
  - The Center for Wound Healing Crozer Chester Medical Center, Chester, Pennsylvania
  - Memorial Hermann Memorial City, Houston, Texas
  - Memorial Hermann South West, Houston, Texas
  - Memorial Hermann South East, Houston, Texas
  - Memorial Hermann Katy Rehab, Katy, Texas
  - Harrison Wound Care & Hyperbaric Medicine, Bremerton, Washington
  - St. Mary's Wound and Hyperbaric Center, Huntington, West Virginia
  - The Center for Wound Healing Cabell Huntington Hospital, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No